CLINICAL TRIAL: NCT00351741
Title: BEST (Burn Center Evaluation of Standard Therapies) Ventilator Mode Study: A Prospective Randomized Controlled Trial
Brief Title: BEST (Burn Center Evaluation of Standard Therapies) Ventilator Mode Study-
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elsa Coates, Administrator, United States Army Institute of Surgical Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-06-005
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Results first posted 2010-12-28 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Burns
Keywords: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Frequency (Experimental): Provide standard ventilatory support for burn patients utilizing high frequency percussive ventilation
  Interventions: Device: Ventilation - High Frequency Percussive Ventilation
- Conventional (Active Comparator): Standard ventilator support for non burned patients utilizing lung protective low tidal volume ventilation
  Interventions: Device: Ventilation - ARDSnet

INTERVENTIONS:
Device: Ventilation - High Frequency Percussive Ventilation — Ventilatory support delivering high frequency percussive ventilation using the Volumetric Diffusive Respirator
  Other Names: High Frequency Percussive Ventilation; Volumetric Diffusive Respirator
  Arms: High Frequency
Device: Ventilation - ARDSnet — Respiratory support with a conventional mode of ventilation using a conventional ventilator (Draeger Evita XL)
  Other Names: Lung Protective Ventilation; Low Tidal Volume Strategy; Conventional Mechanical Ventilation
  Arms: Conventional

SUMMARY:
The purpose of this study is to compare High Frequency Pressure Ventilation (HFPV) to conventional mechanical ventilation.

Hypothesis: Patients placed on HFPV will have significantly higher number of ventilator-free days compared to patients placed on a conventional volume mode.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled trial comparing HFPV to conventional ventilator modes in the support of burn patients with respiratory failure. Burn patients who develop the need for mechanical ventilation present a variety of challenges that call for innovative therapeutic options. Even in the absence of smoke inhalation injury,decreased chest wall compliance from full thickness burns as well as massive fluid requirements are just a few variables that make it difficult to achieve gas exchange goals when attempting to apply conventional lung protective strategies recommended by the ARDS Net investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are deemed to require ventilatory support for more than 24 hours from the time of screening.

Exclusion Criteria:

* Anticipated extubation within 24 hours of screening
* Patients who are pregnant Patients not expected to survive for more than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin K Chung, MD, Principal Investigator — United States Army Insitute of Surgical Research
Locations (1):
- United States Army Institute of Surgical Research, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Salim A, Martin M. High-frequency percussive ventilation. Crit Care Med. 2005 Mar;33(3 Suppl):S241-5. doi: 10.1097/01.ccm.0000155921.32083.ce. PMID 15753734
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Derived] Chung KK, Wolf SE, Renz EM, Allan PF, Aden JK, Merrill GA, Shelhamer MC, King BT, White CE, Bell DG, Schwacha MG, Wanek SM, Wade CE, Holcomb JB, Blackbourne LH, Cancio LC. High-frequency percussive ventilation and low tidal volume ventilation in burns: a randomized controlled trial. Crit Care Med. 2010 Oct;38(10):1970-7. doi: 10.1097/CCM.0b013e3181eb9d0b. PMID 20639746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After 3 yrs of enrollment, interim analysis revealed a significant number of subjects in the LTV arm required rescue, which served as the trigger to close the study to further enrollment. Between April 2006 and May 2009, 387 patients were screened for eligibility. 155 patients met criteria of which 62 were randomized, 31 in each arm.
Groups:
- High Frequency: Intervention with high frequency percussive ventilation
- Conventional: Low-tidal volume ventilation
Period: Overall Study
Arm/Group | High Frequency | Conventional
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Frequency | Conventional | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (18) | 37 (18) | 36 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 27 | 26 | 53
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Ventilator-free Days During the First 28 Days
Description: The primary end point was ventilator-free days in the first 28 days, defined as the number of days after randomization from day 0 to day 28 alive without ventilator assistance for at least 48 consecutive hrs.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | High Frequency | Conventional
Number analyzed (Participants) | 31 | 31
Days | 12 (9) | 11 (9)

2. Secondary Outcome: Days Free From Nonpulmonary Organ Failure
Description: days free from nonpulmonary organ failure as adapted from the ARDSnet study in the first 28 days.
Time Frame: 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | High Frequency | Conventional
Number analyzed (Participants) | 31 | 31
Days | 15 (11) | 15 (10)

3. Secondary Outcome: Death
Description: In-hospital death.
Time Frame: during hospitalization
Measure: Number; unit: Participants
Arm/Group | High Frequency | Conventional
Number analyzed (Participants) | 31 | 31
Participants | 6 | 6

4. Secondary Outcome: Ventilator Associated Pneumonia
Description: Those who develop both clinical and microscopic evidence of pulmonary infection while on the ventilator.
Time Frame: 28 days
Measure: Number; unit: Participants
Arm/Group | High Frequency | Conventional
Number analyzed (Participants) | 31 | 31
Participants | 10 | 16

5. Secondary Outcome: Need for Rescue Ventilator
Description: Subjects who did not meet predetermined oxygenation and ventilation goals on the study mode despite ventilator- specific optimization were switched to a rescue mode of ventilation.
Time Frame: 28 days
Measure: Number; unit: Participants
Arm/Group | High Frequency | Conventional
Number analyzed (Participants) | 31 | 31
Participants | 2 | 9

6. Secondary Outcome: Barotrauma
Description: Defined as a new pneumothorax, pneumomediastinum, subcutaneous emphysema, interstitial emphysema, or pneumatocele >2 cm in diameter not associated with a vascular procedure, lung biopsy, or thoracentesis.
Time Frame: 28 days
Measure: Number; unit: Participants
Arm/Group | High Frequency | Conventional
Number analyzed (Participants) | 31 | 31
Participants | 0 | 4

7. Secondary Outcome: Ventilator Associated Tracheobronchitis (VATB)
Description: Defined as carinal or mainstem airway friability and sloughing with associated bleeding. Only diagnosed after the patient had spent at least 7 days on the assigned ventilator mode and had not been diagnosed with inhalation injury on admission
Time Frame: checked daily
Measure: Number; unit: Participants
Arm/Group | High Frequency | Conventional
Number analyzed (Participants) | 31 | 31
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Description: Ventilator Associated Pneumonia
Arm/Group | High Frequency | Conventional
Serious Adverse Events (participants affected / at risk) | 10/31 | 16/31
Other Adverse Events (participants affected / at risk) | 2/31 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Frequency (N=31) | Conventional (N=31)
Barotrauma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) — defined as a new pneumothorax, pneumomediastinum,subcutaneous emphysema, interstitial emphysema, or pneumatocele >2 cm in diameter not associated with a vascular procedure, lung biopsy, or thoracentesis.
Ventilator Associtated Pneumonia (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 16 (16) — VAP as defined by the American Thoracic Society and the Infectious Disease Society of America
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Frequency (N=31) | Conventional (N=31)
Ventilator Associated Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Defined as carinal or mainstem airway friability and sloughing with associated bleeding.

LIMITATIONS AND CAVEATS:
After 3 yrs of enrollment, interim analysis revealed a significant number of subjects in the Conventional arm required rescue, which served as the trigger to close the study to further enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No